CLINICAL TRIAL: NCT01356706
Title: Minimally Invasive Liver Surgery for Metastases From Colorectal Cancer: Oncologic Outcome and Prognostic Factors
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Baki Topal, Professor of Surgery, University Hospital, Gasthuisberg
Other Study IDs: CRLM-MILS
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Long-term Oncologic Outcome of MILS in Patients With CRLM and Prognostic Indicators
Keywords: liver metastases; colorectal cancer; surgery; prognosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples for histopathology diagnosis & staging
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRLM: patients with colorectal liver metastases (CRLM) who undergo their primary surgery at UZ. Leuven (single-center academic study)

SUMMARY:
Only few reports exist on long-term survival after minimally invasive liver surgery (MILS for colorectal liver metastases. No data are available assessing prognostic factors in the era of current modern treatment strategies. The aim of the current study is to analyze the long-term oncologic outcome after MILS for metastases from colorectal cancer and determine prognostic indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRLM
* Surgery: resection and/or ablation
* preoperative chemotherapy and/or biological agents are allowed
* postoperative chemotherapy and/or biological agents are allowed
* simultaneous colorectal resection is allowed

Exclusion Criteria:

* primary liver cancer
* benign liver tumors
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients sufering from colorectal liever metastases (CRLM) who undergo minimally invasive liver surgery (MILS) or open liver surgery (OLS)
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2002-10; Primary Completion 2008-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
prognostic variables | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven KUL, Leuven, Vlaams-Brabant, Belgium